CLINICAL TRIAL: NCT04999124
Title: Study of the Characteristics of Non-Alcoholic Fatty Liver Disease (NAFLD) in Type 2 Diabetes Mellitus Patients Followed in a Hospital Environment in Flanders, Belgium
Brief Title: Characteristics of NAFLD Among Type 2 Diabetes Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Mathieu Struyve, Principal Investigator, Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: NaDiA-01
Record Dates: First submitted 2020-11-26; First posted 2021-08-10 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Type2 Diabetes
Keywords: NAFLD; NAFLD, characteristics; type 2 diabetes; hospital
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2 | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Type 2 Diabetes Mellitus patients (Other)
  Interventions: Other: Screening and studying characteristics

INTERVENTIONS:
Other: Screening and studying characteristics — Type 2 diabetes patients have a high risk of developing NAFLD. This was confirmed during previous research, a high prevalence of NAFLD among type 2 diabetes mellitus patients was found. Now we want to determine the characteristics of this population.

SUMMARY:
Type 2 diabetes patients have a high risk of developing NAFLD. This was confirmed during previous research, a high prevalence of NAFLD among type 2 diabetes mellitus patients was found. The investigators want to determine the characteristics of this population.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years,
* having type 2 diabetes,
* able to understand Dutch,
* able to understand the informed consent

Exclusion Criteria:

* excessive alcohol abuse,
* other liver disease,
* secondary causes of steatosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
VCTEM (KPa) measure | up to year four
  The FibroScan® device measures vibration controlled transient elastography (VCTE) (kPa) Based on these values the liver stiffness status will be determined.
CAPTM (dB/m) measure | up to year four
  The FibroScan® device measures controlled attenuation parameter (CAP) (dB/m) Based on these values the liver steatosis status will be determined.
Liver Ultrasound | up to year four
  Out of the EPF (Electronic Patient file) the results of a possible earlier ultrasound are noted in the CRF. The results are noted as 'liver steatosis found' with yes/no answer and the year in which this ultrasound was performed.
Liver biopsy | up to year four
  Out of the EPF the results of a possible earlier ultrasound or liver biopsy are noted in the CRF. The results are noted as previous NAFLD diagnosis with yes/no answer and if confirmed by liver biopsy results. Next the NAS CRN (histological) score is noted.The score ranges from 0-8 and is composed of the unweighted sum of steatosis, ballooning, and lobular inflammation. A score between 0-2 corresponds to no NASH, 3-4 is borderline NASH, and definite NASH has a score between 5 and 8.
Aspartate transaminase (AST) | up to year four
  Out of the EPF the blood parameter AST (U/L) will be collected
Alanine transaminase (ALT) | up to year four
  Out of the EPF the blood parameter ALT (U/L) will be collected.
Gamma glutamyltransferase (GGT) | up to year four
  Out of the EPF the blood parameter GGT (U/L) will be collected.
Lactate dehydrogenase (LDH) | up to year four
  Out of the EPF the blood parameter LDH (U/L) will be collected.
total protein | up to year four
  Out of the EPF the blood parameter total protein (g/L) will be collected.
Albumin | up to year four
  Out of the EPF the blood parameter albumin (mg/dL) will be collected.
Ferritin | up to year four
  Out of the EPF the blood parameter ferritin (µg/L) will be collected.
bilirubin total | up to year four
  Out of the EPF the blood parameter bilirubin total (mg/dL) will be collected.
Exclusion of other liver diseases | up to year four
  hepatitis B, hepatitis C, autoimmune hepatitis, primary biliary cirrhosis, hemochromatosis, Wilson disease and alpha 1 antitrypsin deficiency. NAFLD is a disease of exclusion and therefore the abovementioned parameters are determined out of the EPF.
Weight | up to year four
  The weight (kg)
Height | up to year four
  The height (m)
BMI (Body Mass Index) | up to year four
  The weight (kg) and height (m) will be determined and from this the BMI (kg/m²) will be calculated.
waist circumference | up to year four
  The waist circumference will be measured and noted in cm.
Wellbeing - BAECKE | up to year four
  This questionnaire will be used to estimate the level of physical activity. It exists out of 16 questions about work, sports and leisure time. A higher score means that the person is more active at work, does more sport and has a more active leisure time. Minimum value is 3 and maximum value is 15.
Wellbeing - GAD-7 | up to year four
  General Anxiety Disorder (GAD-7) questionnaire will be used to determine the presence of possible clinically significant anxiety disorder.A higher scores indicates having anxiety. Minimum score is 0 and maximum score is 21.
Wellbeing - PHQ-9 | up to year four
  Patient Health Questionnaire-9 (PHQ-9) will be used to quantify depression symptoms and monitor severity. . Minimum score is 0 and maximum score is 27. A higher score indicates having a depression.
Wellbeing - WPAI-SHP | up to year four
  Workers Productivity and Activity Impairment (WPAI-SHP) questionnaire. By means of 6 questions about work productivity and activity it can be determined if there is absence, productivity loss or a decrease in activities at work. By means of 6 questions about work productivity and activity it can be determined if there is absence, productivity loss or a decrease in activities at work. The score is expressed in percentages (0-100). A higher percentage indicates a higher absence from work and a lower productivity.
Wellbeing - SF-36 | up to year four
  Short Form Health Survey-36 will be used to determine the health related quality of life based on 6 different topics: physical functioning, social functioning, role restrictions, mental wellbeing, energy and pain. The score is expressed in percentages (0-100). A higher percentage indicates a better general wellbeing.
Diagnosis Diabetes | up to year four
  The year of diagnosis is asked to the patient (yr).
Diabetes complications | up to year four
  The complications (retinopathy, nephropathy and neuropathy) of diabetes are asked to the patient and gathered out of the EPF. Answer will be yes/no to each of the complications.

SECONDARY OUTCOMES:
concomitant medication | up to year four
  The medication use will be noted in the CRF
serum creatine | up to year four
  serum creatine (mg/dL)
urine creatine | up to year four
  urine creatine (mg/dL)
micro-albumin | up to year four
  micro-albumin (mg/dL)
albumin/creatine ratio | up to year four
  albumin/creatine ratio (mg/g creat)
estimated glomerular filtration rate | up to year four
  estimated glomerular filtration rate (ml/min/1,73m²).
Triglycerides (mg/dL) | up to year four
  Triglycerides (mg/dL) in blood
HDL (mg/dL) | up to year four
  HDL (mg/dL) in blood
LDL cholesterol (mg/dL) | up to year four
  LDL cholesterol (mg/dL) in blood
Total cholesterol (mg/dL). | up to year four
  Total cholesterol (mg/dL) in blood
thrombocytes | up to year four
  thrombocytes (1000/µL) in blood
fasting glucose (mg/dL) | up to year four
  fasting glucose (mg/dL) in blood
partial alpha fetoprotein (AFP) | up to year four
  partial alpha fetoprotein (AFP) in blood
haemoglobin A1c (%) | up to year four
  haemoglobin A1c (%) in blood

CONTACTS AND LOCATIONS:
Overall Officials: Geert Robaeys, prof. dr., Principal Investigator — Hasselt University; Leen Heyens, drs., Study Chair — Hasselt University
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

IPD SHARING:
Plan to Share IPD: No